CLINICAL TRIAL: NCT00427687
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Parallel-Group Study of the Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of AGG-523 Administered Orally to Subjects With Mild to Moderate Osteoarthritis
Brief Title: Study Evaluating AGG-523 in Subjects With Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3189A1-104
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: AGG-523

SUMMARY:
This study will evaluate the effect of AGG-523 administration on biomarkers related to osteoarthritis. Safety and tolerability of AGG-523 will also be assessed.

ELIGIBILITY:
Inclusion:

* Mild to moderate Osteoarthritis of the target knee.
* Subjects must be generally healthy but enrolled with stable chronic illness if well controlled.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The effect of AGG-523 on biomarkers related to osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Anaheim, California
  - Miami, Florida
  - Altoona, Pennsylvania